CLINICAL TRIAL: NCT05874401
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Trilaciclib vs Placebo in Patients With Extensive Stage Small Cell Lung Cancer (ES-SCLC) Receiving Topotecan Chemotherapy
Brief Title: Trilaciclib vs Placebo in Patients With Extensive Stage Small Cell Lung Cancer (ES-SCLC) Receiving Topotecan
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G1T28-211; 2022-502357-34-00 (Other: EU-CTR)
Record Dates: First submitted 2023-04-12; First posted 2023-05-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Extensive-stage Small-cell Lung Cancer
Keywords: myelosuppression; ES-SCLC; chemotherapy-induced myelosuppression; chemotherapy-induced neutropenia; chemotherapy-induced anemia; myeloprotection
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — trilaciclib; Topotecan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² (Experimental): Patients randomized 1:1 to trilaciclib. Patients receive trilaciclib (240 mg/m²) administered once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of trilaciclib on Days 1 to 5, patients receive topotecan (1.5 mg/m²)
  Interventions: Drug: Trilaciclib; Drug: Topotecan
- Placebo + Topotecan 1.5 mg/m² (Placebo Comparator): Patients are randomized 1:1 to placebo. Patients receive placebo administered once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of placebo on Days 1 to 5, patients receive topotecan (1.5 mg/m²).
  Interventions: Drug: Placebo; Drug: Topotecan

INTERVENTIONS:
Drug: Trilaciclib — Participants will receive intravenous trilaciclib infusion
  Other Names: G1T28; CDK 4/6 inhibitor; cyclin-dependent kinase 4/6 inhibitor
  Arms: Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m²
Drug: Placebo — Participants will receive intravenous placebo infusion
  Arms: Placebo + Topotecan 1.5 mg/m²
Drug: Topotecan — Participants will receive intravenous topotecan infusion
  Other Names: Hycamtin

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to assess whether trilaciclib administered prior to topotecan is non-inferior to placebo administered prior to topotecan with regard to overall survival.

DETAILED DESCRIPTION:
The study will include 3 study phases: Screening Phase, Treatment Phase, and Survival Follow-up Phase. Patients randomized in this study will receive trilaciclib/placebo + topotecan 1.5 mg/m2 until disease progression, unacceptable toxicity, withdrawal of consent, Investigator decision to discontinue treatment, or the end of the trial, whichever comes first.

Trilaciclib was approved by the United States (US) Food and Drug Administration (FDA) as a treatment to decrease the incidence of chemotherapy-induced myelosuppression in adult patients when administered prior to a platinum/etoposide-containing regimen or topotecan-containing regimen for ES-SCLC. As a post-marketing requirement, the FDA asked the Sponsor to conduct a study in patients with ES-SCLC undergoing chemotherapy to evaluate survival and disease progression following trilaciclib administration in patients treated with a platinum/etoposide-containing regimen or topotecan-containing regimen with at least 2 years of follow-up. This study is designed to fulfill this requirement.

ELIGIBILITY:
Inclusion Criteria:

1. ES-SCLC with confirmed diagnosis of SCLC by histology or cytology
2. Progression during or after prior first or second line chemotherapy. First-line regimen must have been a platinum-containing combination.
3. Measurable or evaluable disease as defined by RECIST v1.1

Exclusion Criteria:

1. History of topotecan (or other topoisomerase I inhibitor) or trilaciclib treatment for SCLC
2. Any chemotherapy, immunotherapy, biologic, investigational, or hormonal therapy for cancer treatment within 3 weeks, except for adjuvant hormonal therapy for breast cancer and prostate cancer
3. Presence of brain metastases/leptomeningeal disease requiring immediate treatment with radiation therapy or steroids
4. Radiotherapy within 2 weeks
5. History of ILD/pneumonitis
6. History of other malignancies, except for curatively treated solid tumors with no evidence of disease for ≥ 2 years or other NCS cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of randomization until date of death due to any cause for those who died; or date of last contact known as alive for those who survived in the study (censored cases), assessed up to 52 months
  To assess the effect of trilaciclib on OS compared with placebo in patients receiving topotecan

SECONDARY OUTCOMES:
Anti-tumor efficacy | From date of randomization until date of documented radiologic disease progression per RECIST v1.1 or death due to any cause, whichever comes first, assessed up to 52 months
  To assess the effect of trilaciclib on Progression Free Survival (PFS) compared with placebo in patients receiving Topotecan
Anti-tumor efficacy | From date of randomization until the occurrence of progressive disease, withdrawal of consent, or initiation of subsequent anti-cancer therapy, assessed up to 52 months
  To assess the effect of trilaciclib on objective response rate (ORR) compared with placebo in patients receiving Topotecan
Anti-tumor efficacy | From date of first objective response of complete response (CR) or partial response (PR) and the first date that progressive disease is objectively documented or death, whichever comes first, assessed up to 52 months
  To assess the effect of trilaciclib on duration of response (DOR) compared with placebo in patients receiving Topotecan
Neutrophil-related myeloprotection efficacy | From date of randomization until end of cycle 1 (each cycle is 21 days)
  Duration of severe (CTCAE Grade 4) neutropenia in Cycle 1
Neutrophil-related myeloprotection efficacy | From date of randomization until end of treatment, assessed up to 52 months
  Occurrence of severe (CTCAE Grade 4) neutropenia and febrile neutropenia AEs
Neutrophil-related myeloprotection efficacy | From date of randomization until end of treatment, assessed up to 52 months
  Occurrence of G-CSF administration
RBC related myeloprotection efficacy | From date of randomization until end of treatment, assessed up to 52 months
  Occurrence of CTCAE Grade 3 or 4 decreased hemoglobin laboratory values and ESA administration
RBC related myeloprotection efficacy | From date of randomization until end of Week 5
  RBC transfusions on or after Week 5 (occurrence)
RBC related myeloprotection efficacy | From date of randomization until end of Week 5
  RBC transfusions on or after Week 5 (number of transfusions)
Platelet related myeloprotection efficacy | From date of randomization until end of treatment, assessed up to 52 months
  Occurrence of CTCAE Grade 3 or 4 decreased platelet count laboratory values and Platelet transfusions (occurrence)
Platelet related myeloprotection efficacy | From date of randomization until end of treatment, assessed up to 52 months
  Occurrence of CTCAE Grade 3 or 4 decreased platelet count laboratory values and Platelet transfusions (number of transfusions)
Myeloprotection efficacy | From date of randomization until end of treatment, assessed up to 52 months
  Occurrence of hospitalizations due to chemotherapy-induced myelosuppression
Myeloprotection efficacy | From date of randomization until end of treatment, assessed up to 52 months
  Number of hospitalizations due to chemotherapy-induced myelosuppression
Chemotherapy dosing | From the date of randomization until end of treatment, assessed up to 52 months
  To assess the effects of trilaciclib on chemotherapy dosing (delays) compared with placebo when administered prior to topotecan.
Chemotherapy dosing | From the date of randomization until end of treatment, assessed up to 52 months
  To assess the effects of trilaciclib on chemotherapy dosing (reductions) compared with placebo when administered prior to topotecan.
Incidence of Treatment-Emergent Adverse Events as Assessed by CTCAE | From the date of randomization until end of treatment, assessed up to 52 months
  To assess the effects of trilaciclib administered prior to topotecan compared with placebo administered prior to topotecan on occurrence and severity of adverse events by CTCAE, study treatment discontinuation due to adverse events, and trilaciclib adverse events of special interest

CONTACTS AND LOCATIONS:
Overall Officials: Pharmacosmos Clinical and non-clinical Department, Study Director — Pharmacosmos A/S
Locations (1):
- Hospital, Seville, Spain

IPD SHARING:
Plan to Share IPD: No